CLINICAL TRIAL: NCT04868253
Title: Efficacy and Safety of Combination EMB-001 as a Potential Smoking Cessation Treatment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other); Embera NeuroTherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERL-T002
Record Dates: First submitted 2020-10-05; First posted 2021-04-30 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Smoking Cessation; Tobacco Use Disorder
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Metyrapone; Oxazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EMB-001 (Experimental): EMB-001 will be administered utilizing capsules which contain 240 mg of metyrapone and 8 mg of oxazepam (240/8 mg). Subjects will be prescribed 3 capsules (total of 720 mg metyrapone and 24 mg oxazepam) taken twice daily for a total of 12 weeks. After week 12, or if indicated and possibly for a subject who is being discontinued early, subjects will take one capsule of EMB-001, 240/8 mg, twice a day for one additional week (taper dose).
  Interventions: Drug: EMB-01

INTERVENTIONS:
Drug: EMB-01 — EMB-001 is a proprietary combination of metyrapone (a cortisol synthesis inhibitor) and oxazepam (a short to medium acting benzodiazepine).
  Other Names: metyrapone; oxazepam

SUMMARY:
This open-label study will evaluate EMB-001, comprised of metyrapone, a cortisol synthesis inhibitor marketed as a diagnostic drug for testing hypothalamic-pituitary-adrenal (HPA) axis function, combined with oxazepam, an anxiolytic and sedative/hypnotic benzodiazepine, to help smokers abstain from smoking during a 12-week trial period.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the ICF and is able to read and understand the information provided in the ICF.
2. Healthy smokers 21 to 65 years of age (inclusive) at screening.
3. Smokes an average of at least 10 commercially available cigarettes per day for the last 12 months.
4. Has an expired air CO reading of at least 10 ppm at screening.
5. Express a desire to quit smoking within the next 30 days at screening.
6. Serum Cortisol > 3 μg/dL at screening.
7. Willing and able to comply with the requirements of the study.
8. Owns a smart phone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
2. PHQ-9 score greater than 9, or a score greater than 0 on item #9.
3. Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than two times the upper limit of normal or history of liver disease.
4. Have positive serology test results for human immunodeficiency virus (HIV)-1/HIV-2 antibodies, hepatitis B surface antigen, or hepatitis C antibody.
5. High blood pressure (systolic > 150 mmHg or diastolic >95 mmHg) at screening.
6. Body mass index (BMI) less than 18.5 kg/m2 or greater than 35.0 kg/m2.
7. Coronary heart disease, structural cardiac disease, cardiac dysrhythmias, abnormal ECG, syncope, cardiac chest pain, or history of heart attack or heart failure. For males, QTc > 450 msec. For females QTc > 470 msec (using Fridericia correction formula).
8. Has a history of clinically significant drug/alcohol overdose as judged by the Investigator.
9. Has alcohol breathalyzer > 0% at screening.
10. Has a current DSM-5 opioid or benzodiazepine use disorder of any severity or use of these substances or alcohol in amounts that would increase risk of receiving oxazepam as part of EMB-001 or has received psychotherapy or behavioral treatments potentially impacting symptoms of depression, anxiety, or nicotine withdrawal within 30 days of screening, or during the study.
11. Has history of mental illness that, in the opinion of the investigator, may interfere with subject safety or data integrity.
12. Taking antidepressants, CNS or psychoactive medications (e.g., antipsychotics, benzodiazepines, hypnotics) or medications that prolong QTc within the last 30 days of screen or during study.
13. Use of any of these products in the past 30 days:

    1. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, methamphetamines, MDMA (Ecstasy), phencyclidine, benzodiazepines, barbiturates, or opiates at screening);
    2. Experimental (investigational) drugs or biologic;
    3. Chronic opiate use;
    4. Biotin products (Vitamin B7 or B8, Vitamin H, or coenzyme R).
14. Use of glucocorticoids including:

    1. Oral glucocorticoids within 90 days of screen or during study;
    2. Inhaled glucocorticoids within 90 days of screen or during study;
    3. Topical glucocorticoids within 7 days of screen or during the study (except when applied to a small body surface area);
    4. Joint injection within 90 days of screening or during the study.
15. Donation of any blood components within 84 days of screening or during the study or loss of blood ≥ 400 mL within 84 days of screen.
16. Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of enrollment.
17. Pregnant or nursing (by self-report) or has a positive pregnancy test.
18. Female subjects must be of non-childbearing potential. Evidence of non-childbearing potential includes documented surgical sterilization (hysterectomy or bilateral oophorectomy) or being postmenopausal. Postmenopausal is defined clinically as 12 months of amenorrhea in a woman over 45 years of age in the absence of other biological or physiological cause. In addition, women must have a documented serum follicle stimulating hormone (FSH) level > 40 mIU/mL during the Screening Period.
19. Known hypersensitivity to or intolerance of oxazepam, metyrapone, or any benzodiazepine, or severe hypersensitivity reaction (e.g., angioedema) to any drug.
20. Treatment with an investigational drug or biologic within the 30 days preceding the first dose of study medication or plans to take another investigational drug or biologic within 30 days of study completion (including the follow-up visit).
21. Enrollment requirements met.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Smoking Abstinence | Weeks 9 through 12
  Participant self-report of no cigarette smoking (not even a puff).
Smoking Abstinence | 6 month follow-up
  Participant self-report of no cigarette smoking (not even a puff).
Smoking Abstinence | Week 12
  Expired air CO reading of less than 5 ppm

CONTACTS AND LOCATIONS:
Locations (1):
- Rose Research Center, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No